CLINICAL TRIAL: NCT03563833
Title: Investigation of the Effects of Minimal and High Flow Anesthesia on Thiol Disulfide Balance and Peripheral Tissue Saturation (StO2) in Hypotensive Anesthesia Applications
Brief Title: Effects of Minimal and High Flow Anesthesia on Thiol Disulfide Balance and StO2 in Hypotensive Anesthesia Applications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Şule Batçık, Assistant Professor, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2018/64
Record Dates: First submitted 2018-05-20; First posted 2018-06-20 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Oxidative Stress
Keywords: Minimal Flow Anesthesia; Thiol/disulfide balance; Tissue oxygen saturation; hypotensive anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal Flow Anesthesia (Other): Minimal Flow Anesthesia (50% O2, 50% air), Desflurane (MAC = 4,5). In hypotensive anesthesia application; Remifentanil will be used at infusion rates of 0.025-0.1μg / kg / min after a loading dose of 1 μg / kg / min, with mean Arterial Pressure 55-65 mmHg.
  Before the induction of anesthesia and 30 minutes of anesthesia, 2 ml of venous blood sample will be taken from the patients and simultaneous tissue oxygen saturation will be recorded. Serum thiol disulfide levels obtained from the blood sample of the recipient will be studied in the biochemistry research laboratory using the method developed by Erel et al.
  Interventions: Other: Minimal Flow Anesthesia
- High Flow Anesthesia (Other): High Flow Anesthesia (50% O2, 50% air), Desflurane (MAC = 4,5) In hypotensive anesthesia application; Remifentanil will be used at infusion rates of 0.025-0.1μg / kg / min after a loading dose of 1 μg / kg / min, with mean Arterial Pressure 55-65 mmHg.
  Before the induction of anesthesia and 30 minutes of anesthesia, 2 ml of venous blood sample will be taken from the patients and simultaneous tissue oxygen saturation will be recorded. Serum thiol disulfide levels obtained from the blood sample of the recipient will be studied in the biochemistry research laboratory using the method developed by Erel et al.
  Interventions: Other: High Flow Anesthesia

INTERVENTIONS:
Other: Minimal Flow Anesthesia — Minimal Flow Anesthesia with 0,4 L min-1
  Arms: Minimal Flow Anesthesia
Other: High Flow Anesthesia — High Flow Anesthesia with 2 L min-1
  Arms: High Flow Anesthesia

SUMMARY:
The effects of Minimal Flow Anesthesia (0.4 l / min) and High Flow Anaesthesia (2 l / min) on tissue oxygen saturation (St02) and thiol / disulfide balance in hypotensive anesthesia operations will be investigated.

DETAILED DESCRIPTION:
The oxidative stress at the cellular level and the possible effects of general anesthesia techniques on the antioxidant system make the method of anesthesia more important.

The effects of Minimal Flow Anesthesia (0.4 l / min) and High Flow Anaesthesia (2 l / min) on tissue oxygen saturation (St02) and thiol / disulfide balance in hypotensive anesthesia operations will be investigated.

Minimal flow anesthesia is widely used because of its advantages such as cost reduction, prevention of environmental pollution, minimization of heat and humidity loss.

Hypotensive anesthesia is preferred in some specialized surgical procedures in order to reduce bleeding and improve the surgical field of view.

The use of hypotensive anesthesia and inhalation agents may cause hypoperfusion at the tissue level and cause hypoxia-induced oxidative stress and initiate cell damage.

Determining the ideal anesthesia technique in terms of oxidative stress and tissue perfusion will reduce intra- and postoperative risks by protecting patients from the harmful effects of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) I tympanoplasty operations with hypotensive anesthesia,
* ASA (American Society of Anesthesiologists) II tympanoplasty operations with hypotensive anesthesia,

Exclusion Criteria:

* operations in less than one hour
* uncontrolled hypertension
* DM (Diabetes Mellitus)
* cerebrovascular disease
* coagulopathy
* morbid obesity ((BMI ≥ 35)
* renal disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-10-31 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Thiol Disulfide Balance | For two groups; First blood sample will be taken 30 min before the start of surgery, second blood sample will be taken at the 60th min of the surgery
  Change of Oxidative Stress Marker

SECONDARY OUTCOMES:
StO2 | For two groups; simultaneously, 30 min before the start of surgery, 60th min of the surgery
  Change of Peripheral Tissue Oxygen Saturation

CONTACTS AND LOCATIONS:
Overall Officials: Şule Batçık, Asst. Prof., Principal Investigator — Recep Tayyip Erdoğan University Medical School Department of Anesthesia
Locations (1):
- Recep Tayyip Erdoğan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No